CLINICAL TRIAL: NCT01320085
Title: A Phase II, Open-label Study to Assess the Safety and Efficacy of Oral MEK162 in Adults With Locally Advanced and Unresectable or Metastatic Malignant Cutaneous Melanoma, Harboring BRAFV600 or NRAS Mutations
Brief Title: A Phase II Study of Single Agent MEK162 in Patients With Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162X2201; C4211001 (Other: Alias Study Number); 2010-023412-13 (EudraCT Number)
Record Dates: First submitted 2011-03-14; First posted 2011-03-22 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: BRAF or NRAS Mutant Metastatic Melanoma
Keywords: Metastatic melanoma,; BRAF-mutant,; NRAS-mutant
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Melanoma | interventions — binimetinib

ARMS (3):
- BRAFV600 mutant, 45mg bid MEK162 (Experimental): BRAFV600 mutant, 45mg bid MEK162
  Interventions: Drug: MEK162
- NRAS mutant, 45mg bid MEK162 (Experimental): NRAS mutant, 45mg bid MEK162
  Interventions: Drug: MEK162
- BRAFV600 mutant, 60mg bid MEK162 (Experimental): BRAFV600 mutant, 60mg bid MEK162
  Interventions: Drug: MEK162

INTERVENTIONS:
Drug: MEK162

SUMMARY:
The study will assess the safety and efficacy of single-agent MEK162 in adult patients with locally advanced and unresectable or metastatic malignant cutaneous melanoma, harboring BRAFV600E or NRAS mutations.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic cutaneous melanoma AJCC Stage IIIB to IV, not potentially curable with surgery
* BRAF or NRAS mutation in tumor tissue
* All patients enrolled should provide sufficient fresh or archival tumor sample at baseline to enable confirmation of BRAF or NRAS mutations and the additional analyses described in the protocol
* Evidence of measurable tumor disease as per RECIST
* WHO performance status of 0-2
* Adequate organ function and laboratory parameters

Exclusion Criteria:

* History or evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO) or any eye condition that would be considered a risk factor for CSR or RVO
* Patients with unstable CNS metastasis
* Prior treatment with a MEK- inhibitor
* Impaired cardiovascular function
* HIV, active Hepatitis B, and/or active Hepatitis C infection
* Pregnant or nursing (lactating) women
* Women of child-bearing potential UNLESS they comply with protocol contraceptive requirements

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-03-24 (Actual); Primary Completion 2014-01-07 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (10):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - OHSU Knight Cancer Institute, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Cancer Care Associates Medical Oncology, Allentown, Pennsylvania
  - St. Luke's Cancer Center - Allentown Campus, Allentown, Pennsylvania
  - Cancer Care Associates Medical Oncology, Bethlehem, Pennsylvania
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - St. Luke's Hospital - Quakertown Campus, Quakertown, Pennsylvania
- Germany (7):
  - LMU Klinikum der Universität, Munich, Bavaria
  - LMU Klinikum der Universität München, München, Bavaria
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitatsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitatsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - SRH Wald-Klinikum Gera GmbH, Gera, Thuringia
  - LMU Klinikum der Universität München, Munich
- Italy (2):
  - Istituto nazionale Per la Ricerca sul Cancro, Genova
  - Istituto Nazionale per lo studio e la cura dei tumori Fondazione Giovanni Pascale, Napoli
- Netherlands (4):
  - Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam, North Holland
  - Slotervaartziekenhuis, Amsterdam, North Holland
- Universitätsspital Zürich, Zürich (de), Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Ascierto PA, Schadendorf D, Berking C, Agarwala SS, van Herpen CM, Queirolo P, Blank CU, Hauschild A, Beck JT, St-Pierre A, Niazi F, Wandel S, Peters M, Zubel A, Dummer R. MEK162 for patients with advanced melanoma harbouring NRAS or Val600 BRAF mutations: a non-randomised, open-label phase 2 study. Lancet Oncol. 2013 Mar;14(3):249-56. doi: 10.1016/S1470-2045(13)70024-X. Epub 2013 Feb 13. PMID 23414587

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included only those participants for whom the presence of a v-raf murine sarcoma viral oncogene homolog B1 (BRAFV600) or Neuroblastoma RAS viral oncogene homolog (NRAS) gene mutation in the tumor tissue was determined.
Groups:
- Binimetinib 45 mg BRAF: Participants with BRAF mutations received an oral dose of 45 milligrams (mg) of binimetinib (3 tablets each of 15 mg) twice daily, for each 28 days treatment cycle until development of unacceptable toxicity, disease progression, treatment discontinuation by participant refusal or investigator's decision whichever occurred first. Participants were followed up to 30 days after last dose of study drug.
- Binimetinib 45 mg NRAS: Participants with NRAS mutations received an oral dose of 45 mg of binimetinib (3 tablets each of 15 mg) twice daily, for each 28 days treatment cycle until development of unacceptable toxicity, disease progression, treatment discontinuation by participant refusal or investigator's decision whichever occurred first. Participants were followed up to 30 days after last dose of study drug.
- Binimetinib 60 mg BRAF: Participants with BRAF mutations received an oral dose of 60 mg of binimetinib (4 tablets each of 15 mg) twice daily, for each 28 days treatment cycle until development of unacceptable toxicity, disease progression, treatment discontinuation by participant refusal or investigator's decision whichever occurred first. Participants were followed up to 30 days after last dose of study drug.
Period: Overall Study
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Started | 41 | 117 | 25
Completed | 0 | 0 | 0
Not Completed | 41 | 117 | 25
Not completed — Disease Progression | 26 | 93 | 17
Not completed — Adverse Event | 12 | 20 | 5
Not completed — Withdrawal by Subject | 2 | 4 | 1
Not completed — Protocol Deviation | 1 | 0 | 1
Not completed — Administrative problems | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF | Total
Number analyzed (Participants) | 41 | 117 | 25 | 183
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (14.59) | 59.6 (13.74) | 51.3 (9.81) | 57.1 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 33 | 17 | 69
  Male | 22 | 84 | 8 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 10 | 0 | 10
  Not Hispanic or Latino | 41 | 107 | 25 | 173
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 41 | 117 | 25 | 183

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Objective response as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.0, was defined as participants with a best overall response of complete response (CR) or partial response (PR), were recorded from date of randomization or date of start of treatment until date of first documentation of progressive disease (PD) or death due to any cause. CR was defined as complete disappearance of all target and non-target lesions, and sustained for at least 4 weeks apart before progression. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR defined as at least 30 percent (%) decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization or date of start of treatment until date of first documentation of PD or death due to any cause, whichever occurred first (maximum duration of up to 33 months)
Population: The full analysis set included all randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 41 | 117 | 25
percentage of participants | 4.9 [0.6 to 16.5] | 14.5 [8.7 to 22.2] | 12.0 [2.5 to 31.2]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS as assessed by investigator per RECIST v1.0, was defined as time (in months) from date of randomization or date of start of treatment to first documentation of PD or date of death due to any cause or data censoring date, whichever occurred first. PD was defined for target disease as at least a 20% increase in sum of longest diameters of all measured target lesions, taking as reference smallest sum on study (this included baseline sum if that was smallest on study), sum also demonstrated absolute increase of greater than or equal to (>=) 5 mm, or appearance of >=1 new lesions. For non-target disease: PD was defined as unequivocal progression of pre-existing lesions and if overall tumor burden increased sufficiently to merit discontinuation of therapy; appearance of any new unequivocal malignant lesion was also considered PD. If a participant did not had an event, data censoring was done at the date of last adequate tumor assessment. Analysis was performed using Kaplan-Meier method.
Time Frame: From date of randomization or date of start of treatment until date of first documentation of PD or date of death due to any cause or date of data censoring, whichever occurred first (maximum duration of up to 33 months)
Population: The full analysis set included all randomized participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 41 | 117 | 25
months | 3.5 [1.9 to 3.8] | 3.6 [2.6 to 3.8] | 1.8 [1.5 to 3.7]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time (in months) from the date of randomization or date of start of treatment to the date of death due to any cause or data censoring date, whichever occurred first. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: From date of randomization or date of start of treatment to date of death due to any cause or date of censoring, whichever occurred first (maximum duration of up to 33 months)
Population: The full analysis set included all randomized participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 41 | 117 | 25
months | NA [NA to NA] — Median, upper limit and lower limit of 95% Confidence Interval (CI) could not be estimated due to less number of participants with event. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI could not be estimated due to less number of participants with event. | 16.6 [4.9 to NA] — The upper limit of 95% CI could not be estimated due to less number of participants with event.

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR:time from first documentation of OR (confirmed CR or PR) to first documentation of PD/death due to any cause/data censoring date,whichever occurred first. As per RECIST v1.0, CR:disappearance of all target(T) and non-target (Non-T) lesions sustained for =>4 weeks. Any pathological lymph nodes(T or non-T) reduced in short axis to <10mm. PR:>=30% decrease in sum of diameters(SOD) of T lesions, taking as reference baseline SOD. PD for T lesions:at least a 20% increase in sum of diameters of T lesions, taking as reference smallest sum on study treatment, with absolute increase of >=5 mm,or appearance of >=1 new lesions.PD for Non-T lesions:unequivocal progression of pre-existing lesions/increase in overall tumor burden leading to discontinuation of therapy/appearance of new unequivocal malignant lesion.Data was censored on date of last adequate tumor assessment for participants without an event,who started new anti-cancer treatment prior to assessment,who missed >=2 tumor assessments.
Time Frame: From first documentation of CR or PR until first documentation of tumor progression or death due to any cause or data censoring date, whichever occurred first (maximum duration of up to 33 months)
Population: The full analysis set included all randomized participants who received at least one dose of study drug. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 2 | 17 | 3
months | 3.6 [3.6 to 3.7] | 4.0 [3.7 to NA] — The upper limit of 95% CI could not be estimated due to less number of participants with event. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI could not be estimated due to less number of participants with event.

5. Secondary Outcome: Time to Response (TTR)
Description: TTR as assessed by investigator according to RECIST v1.0, was defined as the time (in months) from date of randomization or date of start of treatment until first documented response (CR or PR) or data censoring date, whichever occurred first. CR was defined as complete disappearance of all target and non-target lesions sustained for at least 4 weeks apart before progression. Any pathological lymph nodes (whether target or non-target) reduced in short axis to <10 mm. PR was defined as at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Participants who did not achieve a confirmed PR or CR, were censored at last adequate tumor assessment date when they did not progress (including deaths not due to underlying disease) or at maximum follow-up (from study start to study end date) when participant had an event for progression-free survival.
Time Frame: From the date of randomization or date of start of treatment to the first documentation of objective response (CR or PR) or data censoring date, whichever occurred first (maximum duration of up to 33 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 2 | 17 | 3
months | 2.2 [1.8 to 2.5] | 1.9 [1.8 to 3.7] | 1.8 [1.8 to 1.8]

6. Secondary Outcome: Number of Participants With Grade 3 or 4 Treatment-Emergent Adverse Reactions Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.0
Description: Adverse drug reaction (ADR) was any untoward medical occurrence attributed to study drug in participants who received study drug. As per NCI-CTCAE v4.0, Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or non-invasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4:life-threatening consequence, urgent intervention indicated; Grade 5:death related to study drug. Treatment-emergent ADRs are between first dose of study drug and up to 30 days after last dose of study drug, that were absent before treatment or that worsened relative to pretreatment state. Number of participants with any Grade 3 or 4 treatment-emergent ADR were reported in this outcome measure.
Time Frame: Baseline up to 30 days after last dose of study drug (for a maximum duration of up to 11 years, approximately)
Population: Safety analysis set included all participants who had received at least one dose of study drug and had at least one valid post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 41 | 117 | 25
Participants | 19 | 52 | 13

7. Secondary Outcome: Number of Participants With Serious Adverse Reactions
Description: A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying) ; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly, important medical event.
Time Frame: Baseline up to 30 days after last dose of study drug (for a maximum duration of up to 11 years, approximately)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 41 | 117 | 25
Participants | 2 | 12 | 4

8. Secondary Outcome: Number of Participants With Shift From Baseline in Laboratory Parameter Values Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE) Grade, Version 4.0 (Hematology)
Description: Hematology per NCI-CTCAE included, Lymphocyte count decreased-(G1:<0.8, G2:<0.8-0.5, G3:<0.5-0.2, G4:<0.2[*10^9/L]); Lymphocyte count increased-(G2:>4-20, G3:>20[*10^9/L]); Neutrophil count decreased-(G1:<1.5, G2:<1.5-1.0, G3:<1.0-0.5, G4:<0.5[*10^9/L]); Activated partial thromboplastin time prolonged (seconds)-(G1:>1.5*upper limit normal (ULN), G2:>1.5-2.5*ULN, G3:>2.5*ULN); Platelet count decreased-(G1:<75.0, G2:<75.0-50.0, G3:<50.0-25.0, G4:<25.0[*10^9/L]); Fibrinogen decreased-(G1:<1.0-0.75*lower limit normal (LLN), G2:<0.75-0.5*LLN, G3:<0.5-0.25*LLN G4:<0.25*LLN); Anemia-(G1:<LLN-100, G2:<100-80, G3:<80 [g/L], G4:Life-threatening, G5:death); Hemoglobin increased-(G1:>0-2 g/dL above ULN, G2:>2-4 g/dL above ULN, G3:>4 g/dL above ULN); Prothrombin time (INR) increased-(G1:>1-1.5, G2:>1.5-2.5, G3:>2.5[*ULN]); WBC decreased-(G1:<3.0*10^9/L, G2:<3.0-2.0*10^9/L, G3:<2.0-1.0*10^9/L, G4:<1.0*10^9/L); WBC increased-(G3:>100,000/mm3, G4:Clinical manifestations of increase in WBC, G5:death).
Time Frame: Baseline up to 30 days after last dose of study drug (for a maximum duration of up to 11 years, approximately)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 41 | 117 | 25
Participants
  Absolute Lymphocytes decreased: Grade 0 baseline to Grade 0 post-baseline | 28 | 63 | 10
  Absolute Lymphocytes decreased: Grade 0 baseline to Grade 1 post-baseline | 1 | 8 | 1
  Absolute Lymphocytes decreased: Grade 0 baseline to Grade 2 post-baseline | 1 | 7 | 0
  Absolute Lymphocytes decreased: Grade 0 baseline to Grade 3 post-baseline | 0 | 0 | 1
  Absolute Lymphocytes decreased: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Absolute Lymphocytes decreased: Grade 1 baseline to Grade 0 post-baseline | 2 | 6 | 3
  Absolute Lymphocytes decreased: Grade 1 baseline to Grade 1 post-baseline | 3 | 12 | 3
  Absolute Lymphocytes decreased: Grade 1 baseline to Grade 2 post-baseline | 1 | 4 | 1
  Absolute Lymphocytes decreased: Grade 1 baseline to Grade 3 post-baseline | 1 | 0 | 0
  Absolute Lymphocytes decreased: Grade 2 baseline to Grade 0 post-baseline | 1 | 4 | 0
  Absolute Lymphocytes decreased: Grade 2 baseline to Grade 1 post-baseline | 2 | 2 | 0
  Absolute Lymphocytes decreased: Grade 2 baseline to Grade 2 post-baseline | 0 | 4 | 4
  Absolute Lymphocytes decreased: Grade 2 baseline to Grade 3 post-baseline | 0 | 3 | 1
  Absolute Lymphocytes decreased: Grade 3 baseline to Grade 2 post-baseline | 0 | 2 | 0
  Absolute Lymphocytes decreased: Grade 3 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Absolute Lymphocytes decreased: 'Missing' baseline to Grade 0 post-baseline | 0 | 1 | 0
  Absolute Lymphocytes increased: Grade 0 baseline to Grade 0 post-baseline | 36 | 110 | 22
  Absolute Lymphocytes increased: Grade 0 baseline to Grade 2 post-baseline | 4 | 6 | 2
  Absolute Lymphocytes increased: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Absolute Lymphocytes increased: 'Missing' baseline to Grade 0 post-baseline | 0 | 1 | 0
  Absolute Neutrophils (Segmented and Bands): Grade 0 baseline to Grade 0 post-baseline | 38 | 100 | 21
  Absolute Neutrophils (Segmented and Bands): Grade 0 baseline to Grade 1 post-baseline | 0 | 2 | 0
  Absolute Neutrophils (Segmented and Bands): Grade 0 baseline to Grade 3 post-baseline | 0 | 0 | 2
  Absolute Neutrophils (Segmented and Bands): Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Absolute Neutrophils (Segmented and Bands): Grade 1 baseline to Grade 0 post-baseline | 0 | 1 | 0
  Absolute Neutrophils (Segmented and Bands): Grade 1 baseline to Grade 1 post-baseline | 0 | 2 | 0
  Absolute Neutrophils (Segmented and Bands): Grade 1 baseline to Grade 2 post-baseline | 0 | 1 | 0
  Absolute Neutrophils (Segmented and Bands): Grade 1 baseline to Grade 3 post-baseline | 1 | 0 | 0
  Absolute Neutrophils (Segmented and Bands): Grade 2 baseline to Grade 1 post-baseline | 0 | 1 | 0
  Absolute Neutrophils (Segmented and Bands): Grade 2 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Absolute Neutrophils (Segmented and Bands): Grade 3 baseline to Grade 1 post-baseline | 1 | 0 | 0
  Absolute Neutrophils (Segmented and Bands): Grade 3 baseline to Grade 3 post-baseline | 0 | 0 | 1
  Absolute Neutrophils (Segmented and Bands): Grade 4 baseline to Grade 0 post-baseline | 0 | 1 | 0
  Absolute Neutrophils (Segmented and Bands): 'Missing' baseline to Grade 0 post-baseline | 0 | 4 | 0
  Absolute Neutrophils (Segmented and Bands): 'Missing' baseline to 'Missing' post-baseline | 0 | 4 | 0
  Activated partial thromboplastin time: Grade 0 baseline to Grade 0 post-baseline | 31 | 96 | 19
  Activated partial thromboplastin time: Grade 0 baseline to Grade 1 post-baseline | 3 | 14 | 2
  Activated partial thromboplastin time: Grade 0 baseline to Grade 2 post-baseline | 0 | 1 | 1
  Activated partial thromboplastin time: Grade 0 baseline to Grade 3 post-baseline | 1 | 0 | 0
  Activated partial thromboplastin time: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Activated partial thromboplastin time: Grade 1 baseline to Grade 0 post-baseline | 0 | 1 | 0
  Activated partial thromboplastin time: Grade 1 baseline to Grade 1 post-baseline | 1 | 3 | 1
  Activated partial thromboplastin time: Grade 1 baseline to Grade 2 post-baseline | 1 | 1 | 0
  Activated partial thromboplastin time: Grade 2 baseline to Grade 2 post-baseline | 0 | 1 | 0
  Activated partial thromboplastin time: 'Missing' baseline to Grade 0 post-baseline | 2 | 0 | 1
  Activated partial thromboplastin time: 'Missing' baseline to 'Missing' post-baseline | 1 | 0 | 0
  Platelet count (Direct): Grade 0 baseline to Grade 0 post-baseline | 36 | 97 | 21
  Platelet count (Direct): Grade 0 baseline to Grade 1 post-baseline | 2 | 14 | 3
  Platelet count (Direct): Grade 0 baseline to Grade 2 post-baseline | 0 | 1 | 0
  Platelet count (Direct): Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Platelet count (Direct): Grade 1 baseline to Grade 0 post-baseline | 1 | 0 | 0
  Platelet count (Direct): Grade 1 baseline to Grade 1 post-baseline | 0 | 4 | 0
  Platelet count (Direct): Grade 1 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Platelet count (Direct): 'Missing' baseline to Grade 0 post-baseline | 1 | 0 | 0
  Fibrinogen decreased: Grade 0 baseline to Grade 0 post-baseline | 8 | 19 | 8
  Fibrinogen decreased: Grade 0 baseline to Grade 1 post-baseline | 11 | 52 | 6
  Fibrinogen decreased: Grade 0 baseline to Grade 2 post-baseline | 10 | 32 | 7
  Fibrinogen decreased: Grade 0 baseline to Grade 3 post-baseline | 0 | 8 | 2
  Fibrinogen decreased: Grade 0 baseline to Grade 4 post-baseline | 2 | 1 | 0
  Fibrinogen decreased: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Fibrinogen decreased: Grade 2 baseline to Grade 0 post-baseline | 0 | 1 | 0
  Fibrinogen decreased: 'Missing' baseline to Grade 0 post-baseline | 6 | 4 | 1
  Fibrinogen decreased: 'Missing' baseline to 'Missing' post-baseline | 3 | 0 | 0
  Haemoglobin decreased: Grade 0 baseline to Grade 0 post-baseline | 3 | 22 | 7
  Haemoglobin decreased: Grade 0 baseline to Grade 1 post-baseline | 10 | 35 | 4
  Haemoglobin decreased: Grade 0 baseline to Grade 2 post-baseline | 1 | 4 | 1
  Haemoglobin decreased: Grade 0 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Haemoglobin decreased: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Haemoglobin decreased: Grade 1 baseline to Grade 0 post-baseline | 0 | 4 | 1
  Haemoglobin decreased: Grade 1 baseline to Grade 1 post-baseline | 16 | 27 | 6
  Haemoglobin decreased: Grade 1 baseline to Grade 2 post-baseline | 5 | 16 | 4
  Haemoglobin decreased: Grade 1 baseline to Grade 3 post-baseline | 0 | 3 | 1
  Haemoglobin decreased: Grade 2 baseline to Grade 1 post-baseline | 2 | 0 | 0
  Haemoglobin decreased: Grade 2 baseline to Grade 2 post-baseline | 3 | 3 | 0
  Haemoglobin decreased: Grade 2 baseline to Grade 3 post-baseline | 0 | 2 | 0
  Haemoglobin increased: Grade 0 baseline to Grade 0 post-baseline | 40 | 115 | 24
  Haemoglobin increased: Grade 0 baseline to Grade 1 post-baseline | 0 | 2 | 0
  Haemoglobin increased: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Prothrombin time: Grade 0 baseline to Grade 0 post-baseline | 15 | 40 | 11
  Prothrombin time: Grade 0 baseline to Grade 1 post-baseline | 20 | 56 | 9
  Prothrombin time: Grade 0 baseline to Grade 2 post-baseline | 0 | 2 | 1
  Prothrombin time: Grade 0 baseline to Grade 3 post-baseline | 1 | 2 | 0
  Prothrombin time: Grade 0 baseline to 'Missing' post-baseline | 0 | 0 | 1
  Prothrombin time: Grade 1 baseline to Grade 1 post-baseline | 0 | 5 | 0
  Prothrombin time: Grade 1 baseline to Grade 3 post-baseline | 0 | 0 | 1
  Prothrombin time: Grade 2 baseline to Grade 2 post-baseline | 1 | 0 | 0
  Prothrombin time: Grade 2 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Prothrombin time: Grade 3 baseline to Grade 3 post-baseline | 1 | 0 | 0
  Prothrombin time: 'Missing' baseline to Grade 0 post-baseline | 2 | 0 | 1
  Prothrombin time: 'Missing' baseline to 'Missing' post-baseline | 1 | 11 | 1
  WBC (Total) decreased: Grade 0 baseline to Grade 0 post-baseline | 35 | 93 | 20
  WBC (Total) decreased: Grade 0 baseline to Grade 1 post-baseline | 2 | 10 | 1
  WBC (Total) decreased: Grade 0 baseline to Grade 2 post-baseline | 0 | 1 | 0
  WBC (Total) decreased: Grade 0 baseline to Grade 3 post-baseline | 0 | 0 | 1
  WBC (Total) decreased: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  WBC (Total) decreased: Grade 1 baseline to Grade 0 post-baseline | 2 | 4 | 0
  WBC (Total) decreased: Grade 1 baseline to Grade 1 post-baseline | 0 | 5 | 0
  WBC (Total) decreased: Grade 1 baseline to Grade 2 post-baseline | 0 | 1 | 1
  WBC (Total) decreased: Grade 2 baseline to Grade 1 post-baseline | 1 | 2 | 0
  WBC (Total) decreased: Grade 2 baseline to Grade 2 post-baseline | 0 | 1 | 1
  WBC (Total) increased: Grade 0 baseline to Grade 0 post-baseline | 40 | 117 | 24
  WBC (Total)- increased: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1

9. Secondary Outcome: Number of Participants With Shift From Baseline in Laboratory Parameter Values Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE) Grade, Version 4.0 (Chemistries)
Description: Albumin(G1:<30,G2:<30-20,G3:<20[g/L], G4:life-threatening, G5:death);Alkaline phosphatase(G1:>2.5,G2:>2.5-5.0,G3:>5.0-20.0, G4:>20.0[*ULN]);Creatine kinase(G1:>2.5,G2:>2.5-5,G3:>5-10,G4:>10[*ULN]);Creatinine(CT) clearance(G1:<LLN-60,G2:59-30,G3:29-15,G3:<15[ml/min/1.73m^2], G5:death);CT (G1:>1.5,G2:>1.5-3.0,G3:>3.0-6.0,G4:>6.0[*ULN]);Hypomagnesemia(G1:<0.5,G2:<0.5-0.4,G3:<0.4-0.3,G4:<0.3[mmol/L],G5:death);Hypermagnesemia(G1:>1.23,G3:>1.23-3.30, G4:>3.30[mmol/L],G5:death);Hypophosphatemia(G1:<0.8,G2:<0.8-0.6,G3:<0.6-0.3,G4:<0.3[mmol/L], G5:death);Hypokalemia(G1:<3.0,G2:<3.0,G3:<3.0-2.5,G4:<2.5[mmol/L],G5:death);Hyperkalemia(G1:>5.5,G2:>5.5-6.0,G3:>6.0-7.0, G4:>7.0[mmol/L],G5:death);AST(G1:>3.0,G2:>3.0-5.0,G3:>5.0-20.0,G4:>20.0[*ULN]); ALT(G1:>3.0,G2:>3.0-5.0,G3:>5.0-20.0,G4:>20.0[*ULN]);Hyponatremia(G1:<130,G3:<130-120,G4:<120[mmol/L],G5:death);Hypernatremia(G1:150,G2:>150-155,G3:>155-160,G4:>160[mmol/L],G5:death);High blood bilirubin (G1:>1.5,G2:>1.5-3.0,G3:>3.0-10.0,G4:>10.0[*ULN]).
Time Frame: Baseline up to 30 days after last dose of study drug (for a maximum duration of up to 11 years, approximately)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 41 | 117 | 25
Participants
  Albumin: Grade 0 baseline to Grade 0 post-baseline | 14 | 43 | 11
  Albumin: Grade 0 baseline to Grade 1 post-baseline | 13 | 41 | 4
  Albumin: Grade 0 baseline to Grade 2 post-baseline | 4 | 19 | 2
  Albumin: Grade 0 baseline to Grade 3 post-baseline | 0 | 0 | 1
  Albumin: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Albumin: Grade 1 baseline to Grade 1 post-baseline | 0 | 2 | 1
  Albumin: Grade 1 baseline to Grade 2 post-baseline | 4 | 3 | 5
  Albumin: Grade 2 baseline to Grade 0 post-baseline | 1 | 0 | 0
  Albumin: Grade 2 baseline to Grade 2 post-baseline | 1 | 3 | 0
  Albumin: Grade 2 baseline to Grade 3 post-baseline | 2 | 1 | 0
  Albumin: 'Missing' baseline to Grade 0 post-baseline | 0 | 3 | 0
  Albumin: 'Missing' baseline to Grade 1 post-baseline | 1 | 1 | 0
  Albumin: 'Missing' baseline to Grade 2 post-baseline | 0 | 1 | 0
  Alkaline phosphatase, serum: Grade 0 baseline to Grade 0 post-baseline | 0 | 44 | 0
  Alkaline phosphatase, serum: Grade 0 baseline to Grade 1 post-baseline | 0 | 21 | 0
  Alkaline phosphatase, serum: Grade 0 baseline to Grade 2 post-baseline | 0 | 2 | 0
  Alkaline phosphatase, serum: Grade 0 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Alkaline phosphatase, serum: Grade 1 baseline to Grade 0 post-baseline | 0 | 1 | 0
  Alkaline phosphatase, serum: Grade 1 baseline to Grade 1 post-baseline | 0 | 7 | 0
  Alkaline phosphatase, serum: Grade 1 baseline to Grade 2 post-baseline | 0 | 3 | 0
  Alkaline phosphatase, serum: Grade 1 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Alkaline phosphatase, serum: Grade 2 baseline to Grade 1 post-baseline | 0 | 1 | 0
  Alkaline phosphatase, serum: Grade 2 baseline to Grade 2 post-baseline | 0 | 1 | 0
  Alkaline phosphatase, serum: Grade 3 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Alkaline phosphatase, serum: 'Missing' baseline to Grade 0 post-baseline | 0 | 2 | 3
  Alkaline phosphatase, serum: 'Missing' baseline to Grade 1 post-baseline | 0 | 1 | 1
  Alkaline phosphatase, serum: 'Missing' baseline to 'Missing' post-baseline | 41 | 31 | 21
  Creatine Kinase: Grade 0 baseline to Grade 0 post-baseline | 10 | 20 | 3
  Creatine Kinase: Grade 0 baseline to Grade 1 post-baseline | 11 | 34 | 6
  Creatine Kinase: Grade 0 baseline to Grade 2 post-baseline | 6 | 27 | 4
  Creatine Kinase: Grade 0 baseline to Grade 3 post-baseline | 4 | 13 | 6
  Creatine Kinase: Grade 0 baseline to Grade 4 post-baseline | 1 | 9 | 1
  Creatine Kinase: Grade 0 baseline to 'Missing' post-baseline | 2 | 0 | 1
  Creatine Kinase: Grade 1 baseline to Grade 3 post-baseline | 2 | 2 | 0
  Creatine Kinase: Grade 1 baseline to Grade 4 post-baseline | 1 | 2 | 0
  Creatine Kinase: Grade 2 baseline to Grade 1 post-baseline | 0 | 1 | 0
  Creatine Kinase: Grade 2 baseline to Grade 4 post-baseline | 0 | 1 | 0
  Creatine Kinase: Grade 3 baseline to Grade 4 post-baseline | 0 | 0 | 1
  Creatine Kinase: 'Missing' baseline to Grade 1 post-baseline | 2 | 4 | 0
  Creatine Kinase: 'Missing' baseline to Grade 2 post-baseline | 1 | 0 | 2
  Creatine Kinase: 'Missing' baseline to Grade 3 post-baseline | 1 | 3 | 0
  Creatine Kinase: 'Missing' baseline to 'Missing' post-baseline | 0 | 1 | 1
  Creatinine Clearance: Grade 0 baseline to Grade 0 post-baseline | 22 | 57 | 16
  Creatinine Clearance: Grade 0 baseline to Grade 1 post-baseline | 5 | 17 | 4
  Creatinine Clearance: Grade 0 baseline to Grade 2 post-baseline | 2 | 7 | 0
  Creatinine Clearance: Grade 0 baseline to Grade 3 post-baseline | 0 | 1 | 1
  Creatinine Clearance: Grade 0 baseline to Grade 4 post-baseline | 0 | 1 | 0
  Creatinine Clearance: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Creatinine Clearance: Grade 1 baseline to Grade 0 post-baseline | 0 | 1 | 0
  Creatinine Clearance: Grade 1 baseline to Grade 1 post-baseline | 6 | 12 | 0
  Creatinine Clearance: Grade 1 baseline to Grade 2 post-baseline | 1 | 7 | 2
  Creatinine Clearance: Grade 2 baseline to Grade 1 post-baseline | 2 | 0 | 0
  Creatinine Clearance: Grade 2 baseline to Grade 2 post-baseline | 1 | 6 | 0
  Creatinine Clearance: Grade 2 baseline to 'Missing' post-baseline | 1 | 0 | 0
  Creatinine Clearance: 'Missing' baseline to 'Missing' post-baseline | 0 | 8 | 1
  Creatinine: Grade 0 baseline to Grade 0 post-baseline | 9 | 12 | 4
  Creatinine: Grade 0 baseline to Grade 1 post-baseline | 27 | 91 | 16
  Creatinine: Grade 0 baseline to Grade 2 post-baseline | 1 | 9 | 0
  Creatinine: Grade 0 baseline to Grade 3 post-baseline | 0 | 0 | 1
  Creatinine: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Creatinine: Grade 1 baseline to Grade 0 post-baseline | 1 | 0 | 0
  Creatinine: Grade 1 baseline to Grade 1 post-baseline | 1 | 4 | 2
  Creatinine: Grade 1 baseline to Grade 2 post-baseline | 1 | 1 | 1
  Hypomagnesemia: Grade 0 baseline to Grade 0 post-baseline | 30 | 78 | 22
  Hypomagnesemia: Grade 0 baseline to Grade 1 post-baseline | 4 | 21 | 2
  Hypomagnesemia: Grade 0 baseline to Grade 2 post-baseline | 0 | 1 | 0
  Hypomagnesemia: Grade 0 baseline to 'Missing' post-baseline | 2 | 0 | 1
  Hypomagnesemia: Grade 1 baseline to Grade 0 post-baseline | 0 | 1 | 0
  Hypomagnesemia: Grade 1 baseline to Grade 1 post-baseline | 1 | 8 | 0
  Hypomagnesemia: Grade 1 baseline to Grade 2 post-baseline | 0 | 1 | 0
  Hypomagnesemia: 'Missing' baseline to Grade 0 post-baseline | 3 | 5 | 0
  Hypomagnesemia: 'Missing' baseline to Grade 1 post-baseline | 1 | 1 | 0
  Hypomagnesemia: 'Missing' baseline to 'Missing' post-baseline | 0 | 1 | 0
  Hypermagnesemia: Grade 0 baseline to Grade 0 post-baseline | 35 | 108 | 22
  Hypermagnesemia: Grade 0 baseline to Grade 1 post-baseline | 0 | 1 | 2
  Hypermagnesemia: Grade 0 baseline to 'Missing' post-baseline | 2 | 0 | 1
  Hypermagnesemia: Grade 3 baseline to Grade 0 post-baseline | 0 | 1 | 0
  Hypermagnesemia: 'Missing' baseline to Grade 0 post-baseline | 4 | 6 | 0
  Hypermagnesemia: 'Missing' baseline to 'Missing' post-baseline | 0 | 1 | 0
  Hypophosphatemia (Inorganic Phosphorus): Grade 0 baseline to Grade 0 post-baseline | 36 | 79 | 20
  Hypophosphatemia (Inorganic Phosphorus): Grade 0 baseline to Grade 1 post-baseline | 1 | 6 | 0
  Hypophosphatemia (Inorganic Phosphorus): Grade 0 baseline to Grade 2 post-baseline | 0 | 7 | 0
  Hypophosphatemia (Inorganic Phosphorus): Grade 0 baseline to Grade 3 post-baseline | 0 | 4 | 1
  Hypophosphatemia (Inorganic Phosphorus): Grade 0 baseline to 'Missing' post-baseline | 2 | 0 | 1
  Hypophosphatemia (Inorganic Phosphorus): Grade 1 baseline to Grade 0 post-baseline | 1 | 3 | 1
  Hypophosphatemia (Inorganic Phosphorus): Grade 1 baseline to Grade 2 post-baseline | 0 | 1 | 0
  Hypophosphatemia (Inorganic Phosphorus): Grade 2 baseline to Grade 0 post-baseline | 0 | 8 | 1
  Hypophosphatemia (Inorganic Phosphorus): Grade 2 baseline to Grade 2 post-baseline | 0 | 7 | 1
  Hypophosphatemia (Inorganic Phosphorus): Grade 2 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Hypophosphatemia (Inorganic Phosphorus): 'Missing' baseline to Grade 0 post-baseline | 1 | 1 | 0
  Hypokalemia: Grade 0 baseline to Grade 0 post-baseline | 33 | 93 | 18
  Hypokalemia: Grade 0 baseline to Grade 2 post-baseline | 3 | 19 | 6
  Hypokalemia: Grade 0 baseline to Grade 3 post-baseline | 1 | 0 | 0
  Hypokalemia: Grade 0 baseline to Grade 4 post-baseline | 1 | 0 | 0
  Hypokalemia: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Hypokalemia: Grade 2 baseline to Grade 0 post-baseline | 1 | 1 | 0
  Hypokalemia: Grade 2 baseline to Grade 2 post-baseline | 0 | 3 | 0
  Hypokalemia: Grade 2 baseline to Grade 4 post-baseline | 1 | 1 | 0
  Hyperkalemia: Grade 0 baseline to Grade 0 post-baseline | 35 | 104 | 21
  Hyperkalemia: Grade 0 baseline to Grade 1 post-baseline | 3 | 6 | 1
  Hyperkalemia: Grade 0 baseline to Grade 2 post-baseline | 0 | 2 | 1
  Hyperkalemia: Grade 0 baseline to Grade 3 post-baseline | 0 | 0 | 1
  Hyperkalemia: Grade 0 baseline to Grade 4 post-baseline | 0 | 1 | 0
  Hyperkalemia: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Hyperkalemia: Grade 1 baseline to Grade 0 post-baseline | 0 | 4 | 0
  Hyperkalemia: Grade 1 baseline to Grade 1 post-baseline | 1 | 0 | 0
  Hyperkalemia: Grade 2 baseline to Grade 0 post-baseline | 1 | 0 | 0
  AST: Grade 0 baseline to Grade 0 post-baseline | 11 | 33 | 5
  AST: Grade 0 baseline to Grade 1 post-baseline | 24 | 67 | 13
  AST: Grade 0 baseline to Grade 2 post-baseline | 0 | 5 | 1
  AST: Grade 0 baseline to Grade 3 post-baseline | 0 | 1 | 0
  AST: Grade 0 baseline to Grade 4 post-baseline | 0 | 0 | 1
  AST: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  AST: Grade 1 baseline to Grade 0 post-baseline | 1 | 0 | 0
  AST: Grade 1 baseline to Grade 1 post-baseline | 1 | 6 | 3
  AST: Grade 1 baseline to Grade 2 post-baseline | 2 | 2 | 0
  AST: Grade 1 baseline to Grade 3 post-baseline | 0 | 1 | 1
  AST: Grade 2 baseline to Grade 3 post-baseline | 0 | 1 | 0
  AST: Grade 3 baseline to Grade 3 post-baseline | 1 | 0 | 0
  AST: 'Missing' baseline to Grade 1 post-baseline | 0 | 1 | 0
  ALT: Grade 0 baseline to Grade 0 post-baseline | 20 | 58 | 15
  ALT: Grade 0 baseline to Grade 1 post-baseline | 17 | 39 | 5
  ALT: Grade 0 baseline to Grade 2 post-baseline | 0 | 5 | 0
  ALT: Grade 0 baseline to Grade 3 post-baseline | 0 | 1 | 0
  ALT: Grade 0 baseline to Grade 4 post-baseline | 0 | 0 | 1
  ALT: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  ALT: Grade 1 baseline to Grade 0 post-baseline | 0 | 1 | 0
  ALT: Grade 1 baseline to Grade 1 post-baseline | 3 | 7 | 2
  ALT: Grade 1 baseline to Grade 2 post-baseline | 0 | 4 | 1
  ALT: Grade 1 baseline to Grade 3 post-baseline | 0 | 1 | 0
  ALT: Grade 2 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Hyponatremia: Grade 0 baseline to Grade 0 post-baseline | 25 | 92 | 17
  Hyponatremia: Grade 0 baseline to Grade 1 post-baseline | 7 | 11 | 3
  Hyponatremia: Grade 0 baseline to Grade 3 post-baseline | 1 | 5 | 0
  Hyponatremia: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Hyponatremia: Grade 1 baseline to Grade 0 post-baseline | 3 | 5 | 2
  Hyponatremia: Grade 1 baseline to Grade 1 post-baseline | 4 | 2 | 2
  Hyponatremia: Grade 1 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Hyponatremia: Grade 3 baseline to Grade 3 post-baseline | 0 | 1 | 0
  Hypernatremia: Grade 0 baseline to Grade 0 post-baseline | 37 | 101 | 24
  Hypernatremia: Grade 0 baseline to Grade 1 post-baseline | 2 | 14 | 0
  Hypernatremia: Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Hypernatremia: Grade 1 baseline to Grade 0 post-baseline | 1 | 2 | 0
  Bilirubin (total) increased: Grade 0 baseline to Grade 0 post-baseline | 36 | 105 | 22
  Bilirubin (total) increased: Grade 0 baseline to Grade 1 post-baseline | 1 | 7 | 0
  Bilirubin (total) increased: Grade 0 baseline to Grade 2 post-baseline | 0 | 0 | 1
  Bilirubin (total) increased: Grade 0 baseline to Grade 3 post-baseline | 0 | 2 | 0
  Bilirubin (total) increased: Grade 0 baseline to Grade 4 post-baseline | 0 | 1 | 0
  Bilirubin (total) increased: Grade 0 baseline to 'Missing' post-baseline | 2 | 0 | 1
  Bilirubin (total) increased: Grade 1 baseline to Grade 0 post-baseline | 1 | 1 | 1
  Bilirubin (total) increased: Grade 1 baseline to Grade 1 post-baseline | 1 | 1 | 0

10. Secondary Outcome: Number of Participants With Shift From Baseline in Vital Signs Values Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE) Grade, Version 4.0 (Blood Pressure)
Description: Blood pressure included sitting diastolic blood pressure (DBP) and sitting systolic blood pressure (SBP).
Time Frame: Baseline up to 30 days after last dose of study drug (up to maximum of 33 months)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 41 | 117 | 25
Participants
  Sitting SBP (millimeters of mercury): Grade 0 baseline to Grade 0 post-baseline | 4 | 6 | 0
  Sitting SBP (millimeters of mercury): Grade 0 baseline to Grade 1 post-baseline | 7 | 14 | 6
  Sitting SBP (millimeters of mercury): Grade 0 baseline to Grade 2 post-baseline | 1 | 8 | 0
  Sitting SBP (millimeters of mercury): Grade 0 baseline to Grade 3 post-baseline | 0 | 2 | 0
  Sitting SBP (millimeters of mercury): Grade 1 baseline to Grade 0 post-baseline | 2 | 1 | 1
  Sitting SBP (millimeters of mercury): Grade 1 baseline to Grade 1 post-baseline | 10 | 29 | 6
  Sitting SBP (millimeters of mercury): Grade 1 baseline to Grade 2 post-baseline | 7 | 23 | 6
  Sitting SBP (millimeters of mercury): Grade 1 baseline to Grade 3 post-baseline | 2 | 10 | 2
  Sitting SBP (millimeters of mercury): Grade 1 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Sitting SBP (millimeters of mercury): Grade 2 baseline to Grade 1 post-baseline | 0 | 4 | 1
  Sitting SBP (millimeters of mercury): Grade 2 baseline to Grade 2 post-baseline | 3 | 8 | 1
  Sitting SBP (millimeters of mercury): Grade 2 baseline to Grade 3 post-baseline | 2 | 5 | 0
  Sitting SBP (millimeters of mercury): Grade 2 baseline to 'Missing' post-baseline | 1 | 0 | 0
  Sitting SBP (millimeters of mercury): Grade 3 baseline to Grade 2 post-baseline | 0 | 3 | 1
  Sitting SBP (millimeters of mercury): Grade 3 baseline to Grade 3 post-baseline | 1 | 4 | 0
  Sitting DBP (millimeters of mercury): Grade 0 baseline to Grade 0 post-baseline | 9 | 14 | 2
  Sitting DBP (millimeters of mercury): Grade 0 baseline to Grade 1 post-baseline | 7 | 23 | 6
  Sitting DBP (millimeters of mercury): Grade 0 baseline to Grade 2 post-baseline | 5 | 8 | 4
  Sitting DBP (millimeters of mercury): Grade 0 baseline to Grade 3 post-baseline | 3 | 6 | 2
  Sitting DBP (millimeters of mercury): Grade 0 baseline to 'Missing' post-baseline | 1 | 0 | 0
  Sitting DBP (millimeters of mercury): Grade 1 baseline to Grade 0 post-baseline | 1 | 1 | 0
  Sitting DBP (millimeters of mercury): Grade 1 baseline to Grade 1 post-baseline | 5 | 19 | 1
  Sitting DBP (millimeters of mercury): Grade 1 baseline to Grade 2 post-baseline | 5 | 17 | 5
  Sitting DBP (millimeters of mercury): Grade 1 baseline to Grade 3 post-baseline | 1 | 10 | 2
  Sitting DBP (millimeters of mercury): Grade 1 baseline to 'Missing' post-baseline | 1 | 0 | 1
  Sitting DBP (millimeters of mercury): Grade 2 baseline to Grade 0 post-baseline | 0 | 1 | 0
  Sitting DBP (millimeters of mercury): Grade 2 baseline to Grade 1 post-baseline | 0 | 3 | 0
  Sitting DBP (millimeters of mercury): Grade 2 baseline to Grade 2 post-baseline | 1 | 9 | 1
  Sitting DBP (millimeters of mercury): Grade 2 baseline to Grade 3 post-baseline | 1 | 4 | 1
  Sitting DBP (millimeters of mercury): Grade 3 baseline to Grade 2 post-baseline | 0 | 1 | 0
  Sitting DBP (millimeters of mercury): Grade 3 baseline to Grade 3 post-baseline | 1 | 1 | 0

11. Secondary Outcome: Number of Participants With Markedly Abnormal Vital Sign Values: Sitting Pulse Rate
Description: Pre-defined criteria of markedly abnormal vital signs abnormalities was defined as increase or decrease from baseline (>=15 beats per minute) in pulse rate of >=120 beats per minute or less than or equal to (<=) 50 beats per minute.
Time Frame: Baseline up to 30 days after last dose of study drug (up to maximum of 33 months)
Population: Safety analysis set included all participants who had received at least one dose of study drug and had at least one valid post-baseline safety assessment. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 39 | 116 | 24
Participants
  Sitting pulse (High only) (beats per minute) | 1 | 2 | 1
  Sitting pulse (Low only) (beats per minute) | 1 | 6 | 1
  Sitting pulse (High and Low) (beats per minute) | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Markedly Abnormal Vital Sign Values: Weight
Description: Vital signs included assessment of body weight. Body weight (in kilograms) measurements included high and low. Pre-defined criteria of markedly abnormal vital signs abnormalities was defined as increase or decrease from baseline in weight of >=10%.
Time Frame: Baseline up to 30 days after last dose of study drug (up to maximum of 33 months)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 39 | 117 | 24
Participants
  Weight (High) | 6 | 11 | 8
  Weight (Low) | 2 | 8 | 0

13. Secondary Outcome: Number of Participants With Notable Electrocardiogram (ECG) Values
Description: ECG findings included maximum value of >450 millisecond (msec), >480 msec and >500 msec, increase from baseline >30 msec and >60 msec for QT interval corrected using Fridericia's formula (QTcF); maximum value of >450 msec, >480 msec and >500 msec, increase from baseline >30 msec and >60 msec for QT interval corrected using Bazett's formula (QTcB); maximum value of >450 msec, >480 msec and >500 msec, increase from baseline >30 msec and >60 msec for QT interval; RR decrease >25% and to a VR >100, RR increase >25% and to a VR <50 beats per minute for VR interval; an increase >25% and to a value >200 msec for PR interval; an increase >25% and to a value >110 msec for QRS interval.
Time Frame: Baseline up to 30 days after last dose of study drug (up to maximum of 33 months)
Population: Safety analysis set included all participants who had received at least one dose of study drug and had at least one valid post-baseline safety assessment. Here 'number analyzed' signifies participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 41 | 117 | 25
Participants
  QTcF (millisecond): New >450: number analyzed (Participants) | 34 | 104 | 23
  QTcF (millisecond): New >450 | 5 | 15 | 3
  QTcF (millisecond): New >480: number analyzed (Participants) | 37 | 109 | 23
  QTcF (millisecond): New >480 | 1 | 4 | 0
  QTcF (millisecond): New >500: number analyzed (Participants) | 37 | 109 | 23
  QTcF (millisecond): New >500 | 0 | 0 | 0
  QTcF (millisecond): Increase from baseline >30: number analyzed (Participants) | 37 | 109 | 23
  QTcF (millisecond): Increase from baseline >30 | 4 | 24 | 5
  QTcF (millisecond): Increase from baseline >60: number analyzed (Participants) | 37 | 109 | 23
  QTcF (millisecond): Increase from baseline >60 | 1 | 1 | 0
  QTcB (millisecond): New >450: number analyzed (Participants) | 30 | 94 | 21
  QTcB (millisecond): New >450 | 4 | 26 | 6
  QTcB (millisecond): New >480: number analyzed (Participants) | 35 | 108 | 22
  QTcB (millisecond): New >480 | 3 | 7 | 2
  QTcB (millisecond): New >500: number analyzed (Participants) | 37 | 109 | 23
  QTcB (millisecond): New >500 | 0 | 3 | 1
  QTcB (millisecond): Increase from baseline >30: number analyzed (Participants) | 37 | 109 | 23
  QTcB (millisecond): Increase from baseline >30 | 6 | 29 | 6
  QTcB (millisecond): Increase from baseline >60: number analyzed (Participants) | 37 | 109 | 23
  QTcB (millisecond): Increase from baseline >60 | 0 | 2 | 3
  QT (millisecond): New >450: number analyzed (Participants) | 37 | 105 | 23
  QT (millisecond): New >450 | 6 | 13 | 1
  QT (millisecond): New >480: number analyzed (Participants) | 37 | 107 | 23
  QT (millisecond): New >480 | 2 | 4 | 0
  QT (millisecond): New >500: number analyzed (Participants) | 37 | 109 | 23
  QT (millisecond): New >500 | 1 | 1 | 0
  QT (millisecond): Increase from baseline >30: number analyzed (Participants) | 37 | 109 | 23
  QT (millisecond): Increase from baseline >30 | 14 | 54 | 9
  QT (millisecond): Increase from baseline >60: number analyzed (Participants) | 37 | 109 | 23
  QT (millisecond): Increase from baseline >60 | 3 | 13 | 3
  VR (beats per minute): RR decrease >25% & to a VR >100: number analyzed (Participants) | 37 | 109 | 23
  VR (beats per minute): RR decrease >25% & to a VR >100 | 2 | 6 | 2
  VR (beats per minute): RR increase >25% & to a VR <50: number analyzed (Participants) | 37 | 109 | 23
  VR (beats per minute): RR increase >25% & to a VR <50 | 3 | 8 | 2
  PR (millisecond): Increase >25% & to a value >200: number analyzed (Participants) | 36 | 106 | 23
  PR (millisecond): Increase >25% & to a value >200 | 1 | 6 | 0
  QRS (millisecond): Increase >25% & to a value >110: number analyzed (Participants) | 37 | 109 | 23
  QRS (millisecond): Increase >25% & to a value >110 | 1 | 5 | 1

14. Secondary Outcome: Number of Participants With Change From Baseline in Abnormal Ophthalmoscopy Values- by Fundoscopy
Description: Fundoscopy examination included an examination of the retina, vitreous, macula, optic nerve, optic nerve pallor, choroid and other new abnormalities in either or both eyes. New abnormalities were identified where the baseline assessment showed no abnormalities in a particular eye, but at the post-dose time point an abnormality was observed. New abnormalities at any time point were reported and included unscheduled assessments.
Time Frame: Baseline up to 30 days after last dose of study drug (for a maximum duration of up to 33 months)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 41 | 117 | 25
Participants
  Retina: New abnormalities (At any time): number analyzed (Participants) | 38 | 112 | 24
  Retina: New abnormalities (At any time) | 10 | 43 | 13
  Vitreous: New abnormalities (At any time): number analyzed (Participants) | 38 | 112 | 24
  Vitreous: New abnormalities (At any time) | 2 | 4 | 1
  Macula: New abnormalities (At any time): number analyzed (Participants) | 38 | 113 | 24
  Macula: New abnormalities (At any time) | 7 | 39 | 9
  Optic Nerve: New abnormalities (At any time): number analyzed (Participants) | 38 | 113 | 24
  Optic Nerve: New abnormalities (At any time) | 1 | 5 | 1
  Optic Nerve Pallor: New abnormalities (At any time): number analyzed (Participants) | 38 | 112 | 24
  Optic Nerve Pallor: New abnormalities (At any time) | 0 | 2 | 0
  Choroid: New abnormalities (At any time): number analyzed (Participants) | 38 | 112 | 24
  Choroid: New abnormalities (At any time) | 1 | 5 | 2
  Other: New abnormalities (At any time): number analyzed (Participants) | 5 | 14 | 2
  Other: New abnormalities (At any time) | 0 | 6 | 1

15. Secondary Outcome: Number of Participants With Change From Baseline in Abnormal Ophthalmoscopy Values- by Slit Lamp Examination
Description: Slit lamp examination included an examination of the conjunctiva, cornea, iris, lens, anterior chamber, lids and other new abnormalities in either or both eyes. New abnormalities were identified where the baseline assessment showed no abnormalities in a particular eye, but at the post-dose time point an abnormality was observed. New abnormalities at any time point were reported and included unscheduled assessments.
Time Frame: Baseline up to 30 days after last dose of study drug (for a maximum duration of up to 33 months)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 41 | 117 | 25
Participants
  Conjunctiva: New abnormalities (At any time): number analyzed (Participants) | 37 | 112 | 24
  Conjunctiva: New abnormalities (At any time) | 4 | 25 | 7
  Cornea: New abnormalities (At any time): number analyzed (Participants) | 37 | 112 | 24
  Cornea: New abnormalities (At any time) | 3 | 8 | 5
  Iris: New abnormalities (At any time): number analyzed (Participants) | 37 | 112 | 24
  Iris: New abnormalities (At any time) | 0 | 1 | 0
  Lens: New abnormalities (At any time): number analyzed (Participants) | 37 | 112 | 24
  Lens: New abnormalities (At any time) | 5 | 17 | 3
  Anterior chamber: New abnormalities (At any time): number analyzed (Participants) | 36 | 112 | 24
  Anterior chamber: New abnormalities (At any time) | 0 | 1 | 0
  Lids: New abnormalities (At any time): number analyzed (Participants) | 37 | 112 | 24
  Lids: New abnormalities (At any time) | 6 | 25 | 5
  Other: New abnormalities (At any time): number analyzed (Participants) | 2 | 9 | 0
  Other: New abnormalities (At any time) | 1 | 8 |

16. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval at Steady-State (AUCtau) of Binimetinib
Time Frame: Pre-dose (0 hour), 0.5, 1.5, 3, 8 hours on Day 1 and Day 15 of Cycle 1
Population: Pharmacokinetic (PK) analysis set included all participants who had at least one blood sample providing evaluable PK data. Here 'number analyzed' signifies participants with available data for each specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 37 | 105 | 23
hours*nanogram per milliliter
  Cycle 1, Day 1: number analyzed (Participants) | 4 | 3 | 8
  Cycle 1, Day 1 | 1606.73 (42.55) | 1704.80 (20.37) | 1587.47 (42.49)
  Cycle 1, Day 15: number analyzed (Participants) | 1 | 6 | 4
  Cycle 1, Day 15 | 2438.22 (NA) — The geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 2051.70 (32.63) | 2637.48 (22.04)

17. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Binimetinib
Time Frame: Pre-dose (0 hour), 0.5, 1.5, 3, 8 hours on Day 1 and Day 15 of Cycle 1
Population: PK analysis set included all participants who had at least one blood sample providing evaluable PK data. Here 'number analyzed' signifies participants with available data for each specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 37 | 105 | 23
nanogram per milliliter
  Cycle 1, Day 1: number analyzed (Participants) | 12 | 11 | 19
  Cycle 1, Day 1 | 445.8 (45.8) | 471.6 (34.4) | 542.5 (29.6)
  Cycle 1, Day 15: number analyzed (Participants) | 9 | 13 | 20
  Cycle 1, Day 15 | 385.2 (50.1) | 479.7 (41.1) | 531.3 (44.0)

18. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Binimetinib
Time Frame: Pre-dose (0 hour), 0.5, 1.5, 3, 8 hours on Day 1 and Day 15 of Cycle 1
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 37 | 105 | 23
hours
  Cycle 1, Day 1: number analyzed (Participants) | 12 | 11 | 19
  Cycle 1, Day 1 | 0.68 [0.50 to 3.25] | 1.50 [0.50 to 3.00] | 0.75 [0.50 to 7.98]
  Cycle 1, Day 15: number analyzed (Participants) | 9 | 13 | 20
  Cycle 1, Day 15 | 1.50 [0.75 to 3.17] | 1.48 [0.42 to 8.00] | 1.42 [0.00 to 5.17]

19. Secondary Outcome: Area Under the Curve From Time Zero to Time of Last Quantifiable Concentration (AUC0-last) of Binimetinib
Time Frame: Pre-dose (0 hour), 0.5, 1.5, 3, 8 hours on Day 1 and Day 15 of Cycle 1
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 37 | 105 | 23
hours*nanogram per milliliter
  Cycle 1, Day 1: number analyzed (Participants) | 12 | 11 | 19
  Cycle 1, Day 1 | 1318.38 (47.38) | 1447.07 (21.34) | 1622.66 (37.46)
  Cycle 1, Day 15: number analyzed (Participants) | 9 | 13 | 20
  Cycle 1, Day 15 | 1806.28 (40.86) | 1832.06 (30.71) | 2263.46 (39.84)

20. Secondary Outcome: The Last Time Point of the Last Quantifiable Concentration (Tlast) of Binimetinib
Time Frame: Pre-dose (0 hour), 0.5, 1.5, 3, 8 hours on Day 1 and Day 15 of Cycle 1
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 37 | 105 | 23
hours
  Cycle 1, Day 1: number analyzed (Participants) | 12 | 11 | 19
  Cycle 1, Day 1 | 7.23 [3.23 to 8.00] | 7.98 [7.03 to 8.05] | 7.00 [3.00 to 8.28]
  Cycle 1, Day 15: number analyzed (Participants) | 9 | 13 | 20
  Cycle 1, Day 15 | 7.50 [7.00 to 8.17] | 8.00 [7.02 to 8.43] | 7.50 [3.58 to 8.25]

21. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Binimetinib
Description: Ctrough refers to plasma concentration of Binimetinib observed just before treatment administration.
Time Frame: Pre-dose (0 hour) on Day 15 of Cycle 1
Population: PK analysis set included all participants who had at least one blood sample providing evaluable PK data. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 25 | 65 | 20
nanogram per milliliter | 127.0 (69.6) | 102.3 (79.1) | 136.1 (67.2)

22. Secondary Outcome: Apparent Total Body Clearance (CL/F) of Binimetinib
Description: Drug clearance was defined as a quantitative measure of the rate at which a drug substance was removed from the plasma. Clearance obtained after oral dose was influenced by the fraction of the dose absorbed.
Time Frame: Pre-dose (0 hour), 0.5, 1.5, 3, 8 hours on Day 1 and Day 15 of Cycle 1
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 37 | 105 | 23
liter/hour
  Cycle 1, Day 1: number analyzed (Participants) | 4 | 3 | 8
  Cycle 1, Day 1 | 28.01 (46.90) | 26.40 (20.98) | 37.80 (30.48)
  Cycle 1, Day 15: number analyzed (Participants) | 1 | 6 | 4
  Cycle 1, Day 15 | 18.46 (NA) — The geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 20.50 (26.73) | 21.17 (24.18)

23. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval at Steady-State (AUCtau) of Binimetinib's Metabolite
Time Frame: Pre-dose (0 hour), 0.5, 1.5, 3, 8 hours on Day 1 and Day 15 of Cycle 1
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 37 | 105 | 23
hours*nanogram per milliliter
  Cycle 1, Day 1: number analyzed (Participants) | 2 | 2 | 3
  Cycle 1, Day 1 | 257.73 (7.43) | 170.11 (12.96) | 248.82 (18.33)
  Cycle 1, Day 15: number analyzed (Participants) | 0 | 1 | 1
  Cycle 1, Day 15 |  | 253.93 (NA) — The geometric coefficient of variation could not be estimated as only 1 participant was analyzed. | 322.21 (NA) — The geometric coefficient of variation could not be estimated as only 1 participant was analyzed.

24. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Binimetinib's Metabolite
Time Frame: Pre-dose (0 hour), 0.5, 1.5, 3, 8 hours on Day 1 and Day 15 of Cycle 1
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 37 | 105 | 23
nanogram per milliliter
  Cycle 1, Day 1: number analyzed (Participants) | 12 | 11 | 19
  Cycle 1, Day 1 | 56.37 (39.22) | 49.42 (26.49) | 56.71 (47.62)
  Cycle 1, Day 15: number analyzed (Participants) | 9 | 13 | 20
  Cycle 1, Day 15 | 32.31 (78.98) | 33.55 (58.34) | 25.47 (76.76)

25. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Binimetinib's Metabolite
Time Frame: Pre-dose (0 hour), 0.5, 1.5, 3, 8 hours on Day 1 and Day 15 of Cycle 1
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 37 | 105 | 23
hours
  Cycle 1, Day 1: number analyzed (Participants) | 12 | 11 | 19
  Cycle 1, Day 1 | 1.50 [0.50 to 3.25] | 1.50 [0.50 to 3.00] | 1.50 [0.50 to 7.98]
  Cycle 1, Day 15: number analyzed (Participants) | 9 | 13 | 20
  Cycle 1, Day 15 | 2.50 [0.75 to 3.17] | 1.50 [0.50 to 8.00] | 1.50 [0.00 to 8.00]

26. Secondary Outcome: Area Under the Curve From Time Zero to Time of Last Quantifiable Concentration (AUC0-last) of Binimetinib's Metabolite
Time Frame: Pre-dose (0 hour), 0.5, 1.5, 3, 8 hours on Day 1 and Day 15 of Cycle 1
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 37 | 105 | 23
hours*nanogram per milliliter
  Cycle 1, Day 1: number analyzed (Participants) | 12 | 11 | 19
  Cycle 1, Day 1 | 197.29 (46.15) | 181.60 (29.22) | 189.37 (50.78)
  Cycle 1, Day 15: number analyzed (Participants) | 9 | 13 | 20
  Cycle 1, Day 15 | 157.35 (63.36) | 129.13 (62.80) | 87.11 (79.73)

27. Secondary Outcome: The Last Time Point of the Last Quantifiable Concentration (Tlast) of Binimetinib's Metabolite
Time Frame: Pre-dose (0 hour), 0.5, 1.5, 3, 8 hours on Day 1 and Day 15 of Cycle 1
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 37 | 105 | 23
hours
  Cycle 1, Day 1: number analyzed (Participants) | 12 | 11 | 19
  Cycle 1, Day 1 | 7.23 [3.23 to 8.00] | 7.98 [7.03 to 8.05] | 7.00 [3.00 to 8.28]
  Cycle 1, Day 15: number analyzed (Participants) | 9 | 13 | 20
  Cycle 1, Day 15 | 7.50 [7.00 to 8.17] | 8.00 [2.97 to 8.43] | 7.25 [1.42 to 8.25]

28. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Binimetinib's Metabolite
Description: Ctrough refers to plasma concentration of Binimetinib's metabolite observed just before treatment administration.
Time Frame: Pre-dose (0 hour) on Day 15 of Cycle 1
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 25 | 65 | 20
nanogram per milliliter | 12.85 (80.44) | 11.63 (123.41) | 16.10 (104.21)

29. Secondary Outcome: Percent Change From Baseline in Histological Score (H-score) for Phosphorylated Extracellular Signal-Regulated Kinase (pERK) From Tumor Samples of Cytoplasmic and Nuclear Cellular Compartment
Description: Percent change from baseline in H-score for pERK from tumor samples was assessed and summarized. The H-score is a method of assessing the extent of nuclear immunoreactivity, applicable to steroid receptors.
Time Frame: Baseline up to maximum duration of up to 33 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 3 | 8 | 4
percent change
  Cytoplasmic: Percent change from baseline | -10.90 (26.460) | -50.11 (22.576) | -9.85 (59.566)
  Nuclear: Percent change from baseline | 195.19 (219.585) | -66.83 (47.524) | -32.35 (83.258)

30. Secondary Outcome: Percent Change From Baseline in Delta CT Values for Dual Specificity Phosphatase 6 (DUSP6) Expression From Tumor Samples
Description: The percentage change in DUSP6 gene expression was derived from the Relative Expression Ratio (RER) computed via the Delta Ct method. DUSP6, a protein coding gene was used as a biomarker of inhibition of the mitogen-activated protein kinase (MEK) pathway.
Time Frame: Baseline up to maximum duration of up to 33 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
Number analyzed (Participants) | 3 | 8 | 3
percent change | -50.25 (12.069) | -30.82 (42.836) | 29.48 (73.145)

ADVERSE EVENTS:
Time Frame: From baseline up to 30 days after last dose (for a maximum duration of up to 11 years, approximately)
Description: Same event may appear as both an AE and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety set.
Arm/Group | Binimetinib 45 mg BRAF | Binimetinib 45 mg NRAS | Binimetinib 60 mg BRAF
All-Cause Mortality (participants affected / at risk) | 5/41 | 51/117 | 10/25
Serious Adverse Events (participants affected / at risk) | 11/41 | 39/117 | 9/25
Other Adverse Events (participants affected / at risk) | 40/41 | 117/117 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Binimetinib 45 mg BRAF (N=41) | Binimetinib 45 mg NRAS (N=117) | Binimetinib 60 mg BRAF (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0
Retinopathy (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Face oedema (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 3 | 1
Malaise (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 5 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1
Heart rate irregular (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Binimetinib 45 mg BRAF (N=41) | Binimetinib 45 mg NRAS (N=117) | Binimetinib 60 mg BRAF (N=25)
Anaemia (Blood and lymphatic system disorders) | 4 | 17 | 3
Chorioretinopathy (Eye disorders) | 0 | 16 | 1
Diarrhoea (Gastrointestinal disorders) | 18 | 57 | 13
Nausea (Gastrointestinal disorders) | 10 | 37 | 12
Vomiting (Gastrointestinal disorders) | 4 | 21 | 10
Constipation (Gastrointestinal disorders) | 3 | 23 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 13 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 9 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 7 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 9 | 1
Oedema peripheral (General disorders) | 17 | 60 | 14
Fatigue (General disorders) | 12 | 40 | 12
Pyrexia (General disorders) | 5 | 18 | 2
Face oedema (General disorders) | 5 | 11 | 5
Asthenia (General disorders) | 2 | 10 | 0
Rash pustular (Infections and infestations) | 0 | 11 | 2
Blood creatine phosphokinase increased (Investigations) | 12 | 60 | 14
Aspartate aminotransferase increased (Investigations) | 2 | 20 | 2
Alanine aminotransferase increased (Investigations) | 1 | 18 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 10 | 3
Ejection fraction decreased (Investigations) | 0 | 10 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 19 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 9 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 13 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 14 | 2
Dysgeusia (Nervous system disorders) | 9 | 8 | 1
Headache (Nervous system disorders) | 3 | 7 | 4
Dizziness (Nervous system disorders) | 3 | 6 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 15 | 64 | 8
Rash (Skin and subcutaneous tissue disorders) | 16 | 25 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 21 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 18 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 15 | 2
Erythema (Skin and subcutaneous tissue disorders) | 4 | 8 | 3
Hypertension (Vascular disorders) | 2 | 25 | 6
Weight decreased (Investigations) | 2 | 8 | 0
Visual field defect (Nervous system disorders) | 1 | 8 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 6 | 3
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 5 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1 | 0
Defect conduction intraventricular (Cardiac disorders) | 0 | 2 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 5 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Cleft lip (Congenital, familial and genetic disorders) | 0 | 0 | 1
Colour blindness (Congenital, familial and genetic disorders) | 0 | 2 | 0
Congenital cleft hand (Congenital, familial and genetic disorders) | 0 | 2 | 1
Congenital optic nerve anomaly (Congenital, familial and genetic disorders) | 0 | 1 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 2 | 1
Corneal opacity congenital (Congenital, familial and genetic disorders) | 0 | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0
Macular dystrophy congenital (Congenital, familial and genetic disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Ear swelling (Ear and labyrinth disorders) | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Amblyopia (Eye disorders) | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 4 | 1
Blepharospasm (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 2 | 3 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0
Conjunctival irritation (Eye disorders) | 0 | 1 | 0
Conjunctival oedema (Eye disorders) | 0 | 2 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0
Conjunctivochalasis (Eye disorders) | 0 | 1 | 0
Corneal disorder (Eye disorders) | 0 | 1 | 0
Corneal scar (Eye disorders) | 0 | 0 | 1
Detachment of macular retinal pigment epithelium (Eye disorders) | 0 | 1 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 1 | 8 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 5 | 3
Eczema eyelids (Eye disorders) | 0 | 1 | 0
Extraocular muscle paresis (Eye disorders) | 0 | 1 | 0
Eye allergy (Eye disorders) | 0 | 1 | 0
Eye colour change (Eye disorders) | 0 | 1 | 0
Eye degenerative disorder (Eye disorders) | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0
Eye disorder (Eye disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0
Eye movement disorder (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 1
Eye swelling (Eye disorders) | 0 | 2 | 1
Eyelid disorder (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 6 | 1
Glaucoma (Eye disorders) | 0 | 0 | 2
Lacrimation increased (Eye disorders) | 1 | 2 | 1
Lenticular opacities (Eye disorders) | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 1 | 0
Macular oedema (Eye disorders) | 0 | 4 | 0
Maculopathy (Eye disorders) | 0 | 1 | 0
Meibomianitis (Eye disorders) | 0 | 2 | 0
Ocular discomfort (Eye disorders) | 0 | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 2 | 0
Ocular vascular disorder (Eye disorders) | 0 | 1 | 0
Optic disc haemorrhage (Eye disorders) | 1 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 1
Orbital oedema (Eye disorders) | 0 | 1 | 1
Papilloedema (Eye disorders) | 0 | 1 | 0
Paraneoplastic retinopathy (Eye disorders) | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 3 | 10 | 4
Photophobia (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 1 | 1 | 1
Posterior capsule opacification (Eye disorders) | 0 | 1 | 0
Punctate keratitis (Eye disorders) | 0 | 1 | 0
Retinal cyst (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 2 | 3 | 0
Retinal disorder (Eye disorders) | 0 | 2 | 3
Retinal exudates (Eye disorders) | 1 | 2 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0
Retinal oedema (Eye disorders) | 0 | 1 | 0
Retinal pigment epitheliopathy (Eye disorders) | 0 | 5 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0
Retinopathy (Eye disorders) | 1 | 12 | 9
Retinoschisis (Eye disorders) | 0 | 1 | 0
Subretinal fluid (Eye disorders) | 0 | 8 | 1
Trichiasis (Eye disorders) | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 7 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 2
Visual impairment (Eye disorders) | 1 | 5 | 0
Vitreous detachment (Eye disorders) | 1 | 0 | 0
Vitreous disorder (Eye disorders) | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 2 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 2 | 2
Ascites (Gastrointestinal disorders) | 1 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 5 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 4
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Rectal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 2 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 0
Axillary pain (General disorders) | 0 | 2 | 0
Chest pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 5 | 2
Facial pain (General disorders) | 0 | 2 | 0
Feeling cold (General disorders) | 1 | 4 | 0
Gait disturbance (General disorders) | 0 | 1 | 1
General physical health deterioration (General disorders) | 0 | 3 | 1
Granuloma (General disorders) | 0 | 1 | 0
Hypothermia (General disorders) | 0 | 1 | 0
Inflammation (General disorders) | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 3 | 2
Localised oedema (General disorders) | 0 | 3 | 1
Malaise (General disorders) | 0 | 2 | 0
Mucosal dryness (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 2 | 1
Mucous membrane disorder (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 2 | 1
Oedema (General disorders) | 0 | 4 | 2
Pain (General disorders) | 1 | 2 | 1
Performance status decreased (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 2 | 3 | 2
Swelling (General disorders) | 1 | 0 | 0
Ulcer (General disorders) | 0 | 1 | 0
Xerosis (General disorders) | 1 | 5 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0
Allergy to vaccine (Immune system disorders) | 0 | 1 | 0
Angular cheilitis (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Body tinea (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 4 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 4 | 1
Erysipelas (Infections and infestations) | 1 | 4 | 2
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 3
Influenza (Infections and infestations) | 1 | 5 | 0
Lip infection (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 5 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 1
Orchitis (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 3 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 1
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 3 | 1
Skin infection (Infections and infestations) | 0 | 3 | 2
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 3 | 2
Viral infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Anal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 0
Blood albumin increased (Investigations) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 2 | 1
Blood creatine phosphokinase MB increased (Investigations) | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 6 | 2
Blood fibrinogen increased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 2
Blood magnesium decreased (Investigations) | 0 | 2 | 0
Blood phosphorus decreased (Investigations) | 0 | 3 | 0
Blood phosphorus increased (Investigations) | 0 | 2 | 0
Blood potassium decreased (Investigations) | 0 | 2 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 2 | 0
C-reactive protein increased (Investigations) | 0 | 5 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 2 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 4 | 0
Fibrin D dimer increased (Investigations) | 0 | 4 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 6 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 1
Intraocular pressure increased (Investigations) | 1 | 7 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0
Prothrombin time shortened (Investigations) | 1 | 0 | 0
Sinus rhythm (Investigations) | 0 | 1 | 0
Troponin T increased (Investigations) | 0 | 4 | 0
Weight increased (Investigations) | 3 | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 8 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Hemianopia homonymous (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 1
Neurological symptom (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 3 | 3
Confusional state (Psychiatric disorders) | 0 | 2 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 3 | 0
Dysuria (Renal and urinary disorders) | 0 | 3 | 0
Haematuria (Renal and urinary disorders) | 1 | 4 | 0
Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 2 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal odour (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Chronic pigmented purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cutis laxa (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema weeping (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Milia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 7 | 1
Rash maculovesicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 7 | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin maceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythromelalgia (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 2
Haematoma (Vascular disorders) | 0 | 2 | 0
Hyperanemia (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 2
Lymphoedema (Vascular disorders) | 3 | 3 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 1 | 1
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 2 | 0
Troponin increased (Investigations) | 2 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.